CLINICAL TRIAL: NCT04281498
Title: A Phase II Open-label Study of Combined Ruxolitinib and Enasidenib in Patients With Accelerated/Blast-phase Myeloproliferative Neoplasm or Chronic-phase Myelofibrosis With an IDH2 Mutation
Brief Title: Combined Ruxolitinib and Enasidenib in Patients With Accelerated/Blast-phase Myeloproliferative Neoplasm or Chronic-phase Myelofibrosis With an IDH2 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: Celgene Corporation (Industry); Incyte Corporation (Industry); Myeloproliferative Neoplasms Research Consortium (Unknown); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0548-0008; P01CA108671 (NIH); MPN-RC 119 (Other: Myeloproliferative Neoplasms Research Consortium)
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Accelerated/Blast-phase Myeloproliferative Neoplasm; Chronic-phase Myelofibrosis; IDH2 Mutation
Keywords: Phase II; Myelofibrosis; Therapeutic; Ruxolitinib; Enasidenib; IDH2
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; enasidenib

STUDY DESIGN:
Intervention Model Description: Single Arm open-label Study of Combined Ruxolitinib and Enasidenib in Patients with Accelerated/Blast-phase Myeloproliferative Neoplasm or Chronic-phase Myelofibrosis with an IDH2 Mutation, Simons minimax design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with MPN (Experimental): Ruxolitinib and Enasidenib combination therapy
  Interventions: Drug: Ruxolitinib; Drug: Enasidenib

INTERVENTIONS:
Drug: Ruxolitinib — Patients who are on ruxolitinib will continue their current dose. Patients who are not on ruxolitinib will receive ruxolitinib dosing based on platelet count
Drug: Enasidenib — 50mg -100mg daily

SUMMARY:
The presence of IDH mutation is associated with worse survival in patients with myelofibrosis. Moreover IDH mutations are among the most frequently encountered events in MPNs that have progressed to acute myeloid leukemia. Ruxolitinib, a JAK1/2 inhibitor, and enasidenib an IDH2 inhibitor are effective and tolerable treatments for patients with myelofibrosis (MF) and acute myeloid leukemia (AML), respectively. The study team hypothesize that the combination of these agents in patients with MPN with an IDH2 mutation will improve the overall clinical response to therapy.

DETAILED DESCRIPTION:
At this time, there is no standard medical treatment for MPN-AP/BP and most patients with accelerated and blast phase MPN do not respond well to treatment This is a phase II open-label study to evaluate the safety and efficacy of combined ruxolitinib and enasidenib in patients with accelerated/blast-phase myeloproliferative neoplasm or chronic phase myelofibrosis with high risk features and IDH2 mutation.

Ruxolitinib (Jakafi/Jakavi) is FDA approved for myelofibrosis and was shown to reduce splenomegaly and improve symptoms. Enasidenib is a potent inhibitor of the IDH2 mutant enzyme and is FDA approved for relapsed refractory AML where it showed effectivity.

Pre-clinical studies indicate increased disease mitigating effects with the combination of enasidenib and ruxolitinib.

This study will enroll up to 32 patients. Ruxolitinib and enasidenib will be given orally in 28-day cycles.

ELIGIBILITY:
INCLUSION CRITERIA:

* Subjects must be ≥ 18 years at the time of signing the Informed Consent Form (ICF).
* Understanding and voluntary signing an IRB-approved informed consent form.
* Diagnosis of:

  1. Accelerated-phase (≥ 10% blasts in PB or BM) or blast-phase (≥ 20% blasts in PB or BM) myeloproliferative neoplasm (with history of prior myelofibrosis, polycythemia vera, or essential thrombocythemia)
  2. Previously treated patients with myelofibrosis with persistent disease or progressive disease (persistent or progressive splenomegaly, leukocytosis, anemia, or thrombocytopenia) with intermediate-1 or greater risk disease according to 2013 International Working Group (IWG) criteria, and 4-9% circulating blasts.
* Demonstration of an IDH2 mutation.
* Platelet count > 75,000 X 109/L for chronic phase myelofibrosis patients.
* Prior therapy with either ruxolitinib or enasidenib is permitted, but not a combination of ruxolitinib and enasidenib.
* Patients with chronic phase myelofibrosis on ruxolitinib must be on the drug for at least 3 months and on a stable dose for at least one month.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. ECOG 3 status will be allowed if attributable to MPN.
* Patients must have adequate organ function as demonstrated by the following: a. Direct bilirubin < 2.0mg/dL, unless due to Gilbert's disease or current elevations in direct bilirubin associated with existing enasidenib use. b. Serum creatinine< 2.0 mg/dL. c. ALT and AST ≤ 3x upper limit of normal (unless transaminitis is considered to be related to MF).
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to starting enasidenib and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking enasidenib. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* All study participants must be able to swallow oral medication.
* Ability to adhere to the study visit schedule and all protocol requirements.

EXCLUSION CRITERIA:

* Use of any other standard anti-neoplastic drug or growth factor (e.g., anagrelide, G-CSF, lenalidomide, thalidomide clofarabine) except hydroxyurea or experimental drugs, with the exception of ruxolitinib or enasidenib, less than 14 days or 5-half-lives, whichever is longer, prior to starting study therapy and/or lack of recovery from all toxicity (except for alopecia) from previous therapy to Grade 1 or better.

  a. Patients will be permitted to receive hydroxyurea while on study for up to a total of 3 cycles of combined therapy.
* Known prior clinically relevant hypersensitivity reaction to ruxolitinib or enasidenib.
* Prior therapy with enasidenib in combination with ruxolitinib.
* Concurrent use of strong inducers of CYP3A4 (Rifampin, St. John's Wort, Carbamazepine, Phenytoin) and/or the following strong inhibitors of CYP3A4 (protease inhibitor containing HIV anti-retrovirals, cobicistat, clarithromycin, itraconazole, ketoconazole, nefazodone, and telithromycin) are prohibited. Also prohibited are CYP2C9 substrate medications that have a narrow therapeutic range: phenytoin and warfarin.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form, which places the subject at unacceptable risk if he/she were to participate in the study or which confounds the ability to interpret data from the study.
* Lactating females.
* Active uncontrolled infections.
* Patients with active malignancy of other type than required for this study are not eligible with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received.
* Subject has significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) Class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 28 days prior to the start of study treatment.
* QTc interval (Fridericia's correction [QTcF]) > 450 ms

All inclusion and exclusion criteria will be reviewed by the Investigator or qualified designee to ensure that the patient qualifies for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Ruben Mesa, MD, Study Chair — Mays Cancer Center at UT Health; Ronald Hoffman, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Michal Bar-Natan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (11):
- United States (10):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Taussig Cancer Center Institute, Cleveland, Ohio
  - Mays Cancer Center at UT Health San Antonio, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With MPN
Started | 6
Completed | 3
Not Completed | 3
Not completed — Progression of disease | 1
Not completed — Planned SCT | 1
Not completed — Alternative Treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With MPN
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 74 [58 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Prior Hydroxyurea [Count of Participants; unit: Participants] | 4
Prior Ruxolitinib [Count of Participants; unit: Participants] | 4
Prior Decitabine [Count of Participants; unit: Participants]
  Yes | 1
  No | 4
  Unknown | 1
Total Symptom Score (TSS) [Median (Full Range); unit: units on a scale] — TSS asses via Myelofibrosis Symptom Assessment Form. Full scale from 0-47, higher score indicates worse symptoms.
  units on a scale | 10 [0 to 47]
Platelets [Median (Full Range); unit: cells*10^9/L] | 111.0 [16.0 to 524.0]
Bone marrow % blasts [Median (Full Range); unit: % blast cells in bone marrow] | 12.0 [2.0 to 70.0]
Peripheral blood % blasts [Median (Full Range); unit: % blast cells in peripheral blood] | 14.0 [9.0 to 62.0]
Fibrosis grade [Count of Participants; unit: Participants] — degree of fibrosis in bone marrow
  Participants
    0 None | 1
    1 Mild | 1
    2 Severe | 3
    Not assessed | 1
Patient is transfusion dependent: Red blood cells [Count of Participants; unit: Participants]
  Yes | 3
  Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of MPN Participants With Response
Description: The number of treated accelerated-phase and blast-phase MPN patients (primary cohort) that achieve a best response per 2013 International Working Group (IWG) criteria of either complete response (CR), Partial Response (PR), or complete response with incomplete recovery of counts (CRi), when treated with the combination of ruxolitinib with enasidenib within 6 cycles of combined therapy.
  Complete Response with incomplete recovery of counts (CRi) - complete remission (<5% marrow blasts by morphology) with incomplete count recovery (platelet count <100 x 10^9^/L and/or absolute neutrophil count < 1 x 10^9^/L)
  Complete Response (CR) - full marrow recovery; full count recovery; resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH
  Partial Response (PR) - morphologic remission in the peripheral blood but not necessarily in the bone marrow; resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH
Time Frame: 6 Months
Population: Data for participants with MPN
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With MPN
Number analyzed (Participants) | 5
Participants | 2

2. Secondary Outcome: Number of MPN Participants With Blast Response
Description: The number of treated accelerated-phase and blast-phase MPN patients that achieve complete (CBR) and partial blast response (PBR).
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With MPN
Number analyzed (Participants) | 5
Participants | 3

3. Secondary Outcome: Number of MF-CP Participants With Any Response
Description: The number of treated patients with MF-CP and 4%-9% circulating blasts that achieve complete response (CR) Partial Response (PR), clinical improvement (CI) with the combination of ruxolitinib and enasidenib within 6 cycles of combined therapy.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With MPN
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With MPN
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With MPN (N=6)
Abdominal pain (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With MPN (N=6)
Anemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 2
Neutrophil count decreased (Blood and lymphatic system disorders) | 2
Platelet count decreased (Blood and lymphatic system disorders) | 3
White blood cell decreased (Blood and lymphatic system disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Belching (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 2
Creatinine increased (Investigations) | 2
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema limbs (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 1
Fever (Pyrexia) (General disorders) | 2
Headache (Nervous system disorders) | 3
Heart failure (Cardiac disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER COVID-19 (Infections and infestations) | 1
OTHER Ear lobe pain (Ear and labyrinth disorders) | 1
OTHER early satiety (Gastrointestinal disorders) | 1
OTHER Heartburn (Gastrointestinal disorders) | 1
OTHER Night sweats (General disorders) | 1
OTHER Petechial (Skin and subcutaneous tissue disorders) | 1
OTHER Unspecified contact dermatitis (Skin and subcutaneous tissue disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Vertigo (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT04281498/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT04281498/ICF_001.pdf